CLINICAL TRIAL: NCT02760368
Title: A Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Multicenter Phase III Study of the Efficacy and Safety of Olokizumab in Subjects With Moderately to Severely Active Rheumatoid Arthritis Inadequately Controlled by Methotrexate Therapy
Brief Title: Evaluation of the Effectiveness and Safety of Two Dosing Regimens of Olokizumab (OKZ), Compared to Placebo, in Subjects With Rheumatoid Arthritis (RA) Who Are Taking Methotrexate But Have Active Disease
Acronym: CREDO 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: R-Pharm International, LLC (Industry)
Collaborators: Quintiles, Inc. (Industry); OCT Clinical Trials (Other); Mene Research (Other)
Responsible Party: Sponsor
Organization: R-Pharm (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL04041022; 2014-004719-36 (EudraCT Number)
Record Dates: First submitted 2016-04-29; First posted 2016-05-03 (Estimated); Results first posted 2020-10-30 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Rheumatoid Arthritis
Keywords: moderate Rheumatoid Arthritis; severe Rheumatoid Arthritis; subcutaneous; Olokizumab
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — olokizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1: Olokizumab q4w (Experimental): Olokizumab 64 mg Subcutaneous q4w +placebo+ Methotrexate (oral) in order to maintain the blind, subjects randomized to receive OKZ q4w will receive placebo injections at the alternate q4w interval (e.g., Week 2, Week 6, etc.)
  Interventions: Drug: Olokizumab; Drug: Placebo
- Arm 2: Olokizumab q2w (Experimental): Olokizumab 64 mg Subcutaneous q2w + Methotrexate (oral)
  Interventions: Drug: Olokizumab
- Arm 3: Placebo (Placebo Comparator): Placebo Subcutaneous q2w + Methotrexate (oral)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olokizumab — 160 mg/mL sterile solution for SC injection in a 2 mL clear Type I glass vial
  Arms: Arm 1: Olokizumab q4w; Arm 2: Olokizumab q2w
Drug: Placebo — sodium chloride 0.9% solution supplied in polypropylene plastic ampoules of 10 mL cartons to contain 10 ampoules
  Arms: Arm 1: Olokizumab q4w; Arm 3: Placebo

SUMMARY:
The purpose of this study was to determine how effective and safe the study drug Olokizumab was in patients with Rheumatoid Arthritis (RA) who had been already receiving, but not fully responding to treatment with methotrexate (MTX).

The primary objective of this study was to evaluate the efficacy of olokizumab (OKZ) 64 mg administered subcutaneously (SC) once every 2 weeks (q2w) or once every 4 weeks (q4w) relative to placebo in subjects with moderately to severely active rheumatoid arthritis (RA) inadequately controlled by methotrexate (MTX) therapy.

DETAILED DESCRIPTION:
The goal of this Phase III study was to assess the efficacy, tolerability, and safety of OKZ in subjects with moderately to severely active RA who had responded inadequately to MTX. The primary endpoint of the trial was at Week 12. Olokizumab was expected to reduce the disease activity and improve physical function. The study was expected to provide safety information in a large group of subjects over at least a 24 week period.

The CREDO 1 study included a 4-week Screening Period, a double-blind Treatment Period from Week 0 to Week 24, and a Safety Follow-Up Period from Week 24 to Week 44.

At randomization, a total of 428 eligible subjects were randomly assigned to 1 of 3 treatment groups in a 1:1:1 ratio:

1. OKZ 64 mg q4w: SC injection of OKZ 64 mg q4w (alternating with SC injection of placebo OKZ q4w to maintain blinding) + MTX.
2. OKZ 64 mg q2w: SC injection of OKZ 64 mg q2w + MTX.
3. Placebo: SC injection of placebo q2w + MTX

Throughout the double-blind Treatment Period, all subjects were required to remain on a stable dose of background MTX at 15 to 25 mg/week (or ≥ 10 mg/week if there was documented intolerance to higher doses) with a stable route of administration, and concomitant treatment with folic acid ≥5 mg per week or equivalent is required for all subjects. The last dose of study treatment (OKZ or placebo) was at Week 22 in all groups.

Following Visit 2 (randomization), subjects returned to the study site at least every other week through Week 24 for response and safety assessments as per the study Schedule of Events.

Subjects were classified in terms of their response to study treatment at Week 14, with non-responders defined as subjects in any treatment group who had not improved by at least 20% in both swollen and tender joint counts (66-68 joint assessment). Starting at or as close as possible to Week 14, non-responders were administered sulfasalazine and/or hydroxychloroquine as rescue medication in addition to the assigned treatment.

After completion of the 24-week double-blind Treatment Period, subjects either rolled over into the long-term open-label extension (OLE) study or entered the Safety Follow-Up Period. During the Safety Follow-Up Period, subjects returned for visits +4, +8, and +22 weeks after the last dose of study treatment.

Subjects who discontinued the randomized treatment prematurely were required to come for the End of Treatment (EoT) Visit 2 weeks after the last study treatment administration and then continued with the scheduled study visits as per the Schedule of Events.

The study was conducted at approximately 50 sites across 4 countries globally, which included Russia, Belarus, Turkey, and Bulgaria.

ELIGIBILITY:
Inclusion Criteria:

Subjects may be enrolled in the study only if they meet all of the following criteria:

* Subjects willing and able to sign informed consent
* Subjects must have a diagnosis of adult onset RA classified by ACR/EULAR 2010 revised classification criteria for RA for at least 12 weeks prior to Screening.
* Inadequate response to treatment with MTX for at least 12 weeks prior to Screening at a dose of 15 to 25 mg/week (or ≥10 mg/week if intolerant to higher doses).

  * The dose and means of administering MTX must have been stable for at least 6 weeks prior to Screening.
* Subjects must be willing to take folic acid or equivalent throughout the study
* Subjects must have moderately to severely active RA disease as defined by all of the following:

  * ≥6 tender joints (68 joint count) at Screening and baseline; and
  * ≥6 swollen joints (66 joint count) at Screening and baseline; and
  * CRP above ULN at Screening based on the central laboratory results.

Exclusion Criteria:

* Diagnosis of any other inflammatory arthritis or systemic rheumatic disease (e.g., gout, psoriatic or reactive arthritis, Crohn's disease, Lyme disease, juvenile idiopathic arthritis, or systemic lupus erythematosus). However, subjects could have secondary Sjogren's syndrome or hypothyroidism
* Subjects who were Steinbrocker class IV functional capacity (incapacitated, largely or wholly bed-ridden or confined to a wheelchair, with little or no self-care)
* Prior exposure to any licensed or investigational compound directly or indirectly targeting IL-6 or IL-6R (including tofacitinib or other Janus kinases and spleen tyrosine kinase [SYK] inhibitors)
* Prior treatment with cell-depleting therapies, including anti-CD20 or investigational agents (e.g., CAMPATH, anti-CD4, anti-CD5, anti-CD3, and anti-CD19)
* Prior use of bDMARDs, with the following exception:

  • Subjects who discontinued TNFi therapy due to a reason other than lack of efficacy were allowed to enter the study (TNFi therapy was not to be discontinued to facilitate a subject's participation in the study but should instead have been previously discontinued as part of a subject's medical management of RA). The use of TNFi therapy within the following windows prior to baseline was exclusionary:
  1. 4 weeks for etanercept
  2. 8 weeks for infliximab
  3. 10 weeks for adalimumab, certolizumab, and golimumab
* Use of parenteral and/or intra-articular glucocorticoids within 4 weeks prior to baseline
* Use of oral glucocorticoids greater than 10 mg/day prednisone (or equivalent), or change in dosage within 2 weeks prior to baseline
* Prior documented history of no response to hydroxychloroquine and sulfasalazine
* Prior use of cDMARDs (other than MTX) within the following windows prior to baseline (cDMARDs were not to be discontinued to facilitate a subject's participation in the study, but should instead have been previously discontinued as part of a subject's medical management of RA):

  1. 4 weeks for sulfasalazine, azathioprine, cyclosporine, hydroxychloroquine, chloroquine, gold, penicillamine, minocycline, or doxycycline
  2. 12 weeks for leflunomide unless the subject has completed the following elimination procedure at least 4 weeks prior to baseline: Cholestyramine at a dosage of 8 grams 3 times daily for at least 24 hours, or activated charcoal at a dosage of 50 grams 4 times daily for at least 24 hours
  3. 24 weeks for cyclophosphamide
* Vaccination with live vaccines in the 6 weeks prior to baseline or planned vaccination with live vaccines during the study
* Participation in any other investigational drug study within 30 days or 5 times the terminal half-life of the investigational drug, whichever is longer, prior to baseline
* Other treatments for RA (e.g., Prosorba Device/Column) within 6 months prior to baseline
* Use of intra-articular hyaluronic acid injections within 4 weeks prior to baseline
* Use of non-steroidal anti-inflammatory drugs (NSAIDs) on unstable dose or switching of NSAIDs within 2 weeks prior to baseline
* Previous participation in this study (randomized) or another study of OKZ
* Subjects with acute or chronic viral hepatitis B or C infection as detected by blood tests at Screening (e.g., positive for hepatitis B surface antigen [HBsAg], total hepatitis B core antibody [anti-HBc], or hepatitis C virus antibody [HCV Ab])

  a. Subjects who were positive for hepatitis B surface antibody (anti-HBs), but negative for HBsAg and anti-HBc, were eligible
* Subjects with HIV infection
* Subjects with:

  1. Suspected or confirmed current active TB disease or a history of active TB disease
  2. Close contact (i.e., sharing the same household or other enclosed environment, such as a social gathering place, workplace, or facility, for extended periods during the day) with an individual with active TB within 1.5 years prior to Screening.
* Concurrent malignancy or a history of malignancy within the last 5 years (with the exception of successfully treated carcinoma in situ of the cervix and successfully treated basal cell carcinoma and squamous cell carcinoma not less than 1 year prior to Screening [and no more than 3 excised skin cancers within the last 5 years prior to Screening])
* Subjects with any infection requiring oral antibiotic or antiviral therapy in the 2 weeks prior to Screening or at baseline, injectable anti-infective therapy in the last 4 weeks prior to baseline, or serious or recurrent infection with a history of hospitalization in the 6 months prior to baseline
* Subjects with evidence of disseminated herpes zoster infection, zoster encephalitis, meningitis, or other non-self-limited herpes zoster infections in the 6 months prior to baseline
* Subjects with planned surgery during the study or surgery ≤4 weeks prior to Screening and from which the subject had not fully recovered, as judged by the Investigator
* Subjects with diverticulitis or other symptomatic GI conditions that might predispose the subject to perforations, including subjects with a history of such predisposing conditions (e.g., diverticulitis, GI perforation, or ulcerative colitis)
* Pre-existing central nervous system demyelinating disorders (e.g., multiple sclerosis and optic neuritis)
* History of chronic alcohol or drug abuse as judged by the Investigator
* Female subjects who are pregnant, currently lactating, have lactated within the last 12 weeks, or who were planning to become pregnant during the study or within 6 months of last dose of study treatment
* Female subjects of childbearing potential (unless permanent cessation of menstrual periods, determined retrospectively after a woman had experienced 12 months of natural amenorrhea as defined by the amenorrhea with underlying status [e.g., correlative age] or 6 months of natural amenorrhea with documented serum follicle-stimulating hormone levels >40 mIU/mL and estradiol <20 pg/mL) who were not willing to use a highly effective method of contraception during the study and for at least 6 months after the last administration of study treatment OR Male subjects with partners of childbearing potential not willing to use a highly effective method of contraception during the study and for at least 3 months after the last administration of study treatment;
* Subjects with a known hypersensitivity to any component of the OKZ drug product, or placebo
* Subjects with a known hypersensitivity or contraindication to any component of the rescue medication
* History of severe allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2016-05-19 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — R-Pharm
Locations (40):
- Belarus (2):
  - City Clinical Hospital #1, Minsk
  - Vitebsk Regional Clinical Hospital, Vitebsk
- Bulgaria (4):
  - DCC 'Sv. Pantaleymon' OOD, Pleven
  - UMHAT "Kaspela", EOOD, Plovdiv
  - UMHAT "Sv. Ivan Rilski", EAD, Sofia
  - MC "Synexus - Sofia", EOOD, Sofia
- Russia (34):
  - Regional State Budgetary Healthcare Institution "Barnaul City Hospital #4", Barnaul, Altayskiy Kray
  - SAHI of Kemerovo region "Regional Clinical Hospital for War Veterans", Kemerovo, Kemerovo Oblast
  - Medical Center LLC "Maksimum Zdoroviya", Kemerovo, Kemerovo Oblast
  - Budgetary Healthcare Institution "Kursk Regional Clinical Hospital" of Healthcare Committee of Kursk region, Kursk, Kursk Oblast
  - SPb SBHI "Clinical Rheumatological Hospital #25", Fourth Rheumatology Unit, Saint Petersburg, Leningradskaya Oblast'
  - FSBEI HE "First Moscow State Medical University n.a. I.M. Sechenov of MoH of Russian Federation", UCH #1, Moscow, Moscovskaya Oblast
  - FSBEI HE "FMSMU n.a. I.M. Sechenov of MoH of RF", University Hospital #2, Departament of New Drugs Introduction, Moscow, Moscovskaya Oblast
  - SBEI HPE "First Moscow State Medical University n.a. I.M. Sechenov of MoH of Russian Federation" UCH #3, Moscow, Moscovskaya Oblast
  - State Budgetary Healthcare Institution of Moscow "City Clinical Hospital #1 n.a. Pirogov" Healthcare Departament of Moscow, Moscow, Moscovskaya Oblast
  - State Budgetary Healthcare Institution "City Clinical Hospital # 15 n.a O.M. Filatov" of Moscow Healtheare Department, Moscow, Moscow Oblast
  - SBHI of Moscow "City Clinical Hospital #4 of Moscow Healthcare Departament", Moscow, Moscow Oblast
  - SBHI of Nizhny Novgorod Region "Nizhny Novgorod Regional Clinical Hospital n.a.Semashko", Nizhny Novgorod, Nizhny Novgorod Oblast
  - State Autonomous Healthcare Institution of Novosibirsk region "City Polyclinic #1", Novosibirsk, Novosibirsk Oblast
  - LLC "Clinical Diagnostic Center "Ultramed", Omsk, Omsk Oblast
  - Budgetary Healthcare Institution of Omsk Region "Regional Clinical Hospital", Omsk, Omsk Oblast
  - SBHI of the Republic of Karelia "Republican Hospital named after V.A. Baranov", Petrozavodsk, Republic of Karelia
  - State Budgetary Healthcare Institution "Republican Clinical Hospital n.a. G.G. Kuvatov", Ufa, Respublic of Bashkortostan
  - SBEI HPE "Rostov State Medical University" of Ministry of Health of the Russian Federation, Rostov-on-Don, Rostov Oblast
  - State Healthcare Institution "Regional Clinical Hospital", Saratov, Saratov Oblast
  - SBEI HPE "SSMU n.a. V.I. Razumovsky of MoH of RF", Clinical Hospital n.a. S.R. Mirotvorcev, Therapeutic Departament, Saratov, Saratov Oblast
  - Non-governmental Healtheare Institution "Regional Clinical Hospital at Smolensk station of OJSC "Russian Railways", Smolensk, Smolensk Oblast
  - SBHI of Stavropol Region "Stavropol Regional Clinical Hospital", Stavropol, Stavropol Kray
  - State Budgetary Healthcare Institution of Sverdlovsk Region "Sverdlovsk Regional Clinical Hospital #1", Yekaterinburg, Sverdlovsk Oblast
  - SBEI HPE "Ural State Medical University" of MoH of RF based MBI "Central City Clinical Hospital #6", Yekaterinburg, Sverdlovsk Oblast
  - State Autonomous Healthcare Institution "Republican Clinical Hospital of Ministry of Health of Tatarstan Republic, Kazan', The Republic of Tatarstan
  - State Healthcare Institution of Tula region "Tula Regional Clinical Hospital", Tula, Tulskaya Oblast
  - State Healthcare Institution "Ulyanovsk Regional Clinical Hospital", Ulyanovsk, Ulyanovsk Oblast
  - SBHI of Vladimir Region "Regional Clinical Hospital", Rheumatology Departament, Vladimir, Vladimirskaya Oblast’
  - SBHI "Yaroslavl Regional Clinical Hospital", Rheumatology department, Yaroslavl, Yaroslavl Oblast
  - State Autonomous Helthcare Institution of Yaroslavl region "Clinical Hospital of Emergency Care n.a. Solovyev", Yaroslavl, Yaroslavsakaya Oblast
  - FSBSI "Scientific Research Institute of Rheumatology n.a. V.A. Nasonova", Moscow
  - City Clinical Hospital №5 of Nizhny Novgorod, Nizhny Novgorod
  - Ryazan State Medical University n.a. I.P. Pavlov based on Regional Clinical Cardiology Dispensary, Ryazan
  - SBHI "North-West Federat Medical Research Center n.a. V.A.Almazov" of the Ministry of Healthcare of the Russian Federation, Saint Petersburg

REFERENCES:
- [Derived] Nasonov E, Fatenejad S, Feist E, Ivanova M, Korneva E, Krechikova DG, Maslyanskiy AL, Samsonov M, Stoilov R, Zonova EV, Genovese M. Olokizumab, a monoclonal antibody against interleukin 6, in combination with methotrexate in patients with rheumatoid arthritis inadequately controlled by methotrexate: efficacy and safety results of a randomised controlled phase III study. Ann Rheum Dis. 2022 Apr;81(4):469-479. doi: 10.1136/annrheumdis-2021-219876. Epub 2021 Aug 3. PMID 34344706
- See also: Nasonov E, Fatenejad S, Korneva E, Krechikova D. - Safety and Efficacy of Olokizumab in a Phase III Trial of Patients with Moderately to Severely Active Rheumatoid Arthritis Inadequately Controlled by Methotrexate - CREDO1 Study [abstract]. — http://acrabstracts.org/abstract/safety-and-efficacy-of-olokizumab-in-a-phase-iii-trial-of-patients-with-moderately-to-severely-active-rheumatoid-arthritis-inadequately-controlled-by-methotrexate-credo1-study/
- See also: E. Nasonov, R. Stoilov, T. Tyabut, M. C. Genovese. 2020 OP0021 Olokizumab, Monoclonal Antibody Against IL6, in Patients with Moderately to Severely Active Rheumatoid Arthritis Inadequately Controlled by Methotrexate:Results of Phase III CREDO-1 study — http://scientific.sparx-ip.net/archiveeular/?c=a&searchfor=olokizumab&view=1&item=2020OP0021
- See also: E. Nasonov, M. Ivanova, M. Samsonov, T. Tyabut, M. C. Genovese; 2020 THU0176 Olokizumab Improves Patient Reported Outcomes in Patients with Moderately to Severely Active Rheumatoid Arthritis Inadequately Controlled by Methotrexate: Results CREDO-1 study — http://scientific.sparx-ip.net/archiveeular/?c=a&searchfor=olokizumab&view=1&item=2020THU0176

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was conducted at 42 clinical sites (in Belarus, Bulgaria, Russia,Turkey) between May 2016 and April 2018. 785 patients were included, 357 patients screen-failed, 428 patients were randomized (143 patients in OKZ q2w +MTX group, 142 patients in OKZ q4w +MTX group, 143 patients in Placebo q2w +MTX group). 1 subject was randomized by mistake and didn't receive the study treatment. The primary efficacy analysis set included 428 subjects, and the safety analysis set included 427 subjects.
Groups:
- Arm 1: Olokizumab q4w + Methotrexate: Olokizumab 64 mg Subcutaneous q4w + placebo + Methotrexate (oral)
  64 mg Olokizumab administered subcutaneously once every 4 weeks + placebo in order to maintain the blind, subjects randomized to receive OKZ q4w will receive placebo injections at the alternate q4w interval (e.g., Week 2, Week 6, etc.)+concomitant background therapy (Methotrexate) at a stable dose of 15 to 25 mg/week (or ≥10 mg/week if there is documented intolerance to higher doses) with a stable route of administration (oral, subcutaneous, or intramuscular)
- Arm 2: Olokizumab q2w + Methotrexate: Olokizumab 64 mg Subcutaneous q2w + Methotrexate (oral)
  64 mg Olokizumab administered subcutaneously once every 2 weeks + concomitant background therapy (Methotrexate) at a stable dose of 15 to 25 mg/week (or ≥10 mg/week if there is documented intolerance to higher doses) with a stable route of administration (oral, subcutaneous, or intramuscular)
- Arm 3: Placebo + Methotrexate: Placebo Subcutaneous q2w + Methotrexate (oral)
  Placebo administered subcutaneously once every 2 weeks + concomitant background therapy (Methotrexate) at a stable dose of 15 to 25 mg/week (or ≥10 mg/week if there is documented intolerance to higher doses) with a stable route of administration (oral, subcutaneous, or intramuscular)
Period: Overall Study
Arm/Group | Arm 1: Olokizumab q4w + Methotrexate | Arm 2: Olokizumab q2w + Methotrexate | Arm 3: Placebo + Methotrexate
Started | 142 | 143 | 143
Completed | 134 | 130 | 132
Not Completed | 8 | 13 | 11
Not completed — Withdrawal by Subject | 8 | 12 | 9
Not completed — Screen Failure | 0 | 0 | 1
Not completed — Death | 0 | 1 | 0
Not completed — Withdrawal by Sponsor | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Olokizumab q4w + Methotrexate: Olokizumab 64 mg Subcutaneous q4w +placebo q4w+ Methotrexate (oral)
  Olokizumab q4w: 160 mg/mL sterile solution for SC injection in a 2 mL clear Type I glass vial + placebo (sodium chloride 0.9% solution supplied in polypropylene plastic ampoules of 10 mL cartons to contain 10 ampoules)
- Arm 2: Olokizumab q2w + Methotrexate: Olokizumab 64 mg Subcutaneous q2w + Methotrexate (oral)
  Olokizumab q2w: 160 mg/mL sterile solution for SC injection in a 2 mL clear Type I glass vial
- Arm 3: Placebo q2w + Methotrexate: Placebo Subcutaneous q2w + Methotrexate (oral)
  Placebo q2w: sodium chloride 0.9% solution supplied in polypropylene plastic ampoules of 10 mL cartons to contain 10 ampoules
- Total: Total of all reporting groups
Arm/Group | Arm 1: Olokizumab q4w + Methotrexate | Arm 2: Olokizumab q2w + Methotrexate | Arm 3: Placebo q2w + Methotrexate | Total
Number analyzed (Participants) | 142 | 143 | 143 | 428
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 129 | 125 | 124 | 378
  >=65 years | 13 | 18 | 19 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (12.07) | 52.0 (11.77) | 52.7 (11.29) | 51.3 (11.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 116 | 120 | 354
  Male | 24 | 27 | 23 | 74
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  participants: Asian | 0 | 0 | 1 | 1
  participants: Black or African American | 0 | 0 | 0 | 0
  participants: White | 142 | 143 | 142 | 427
  participants: Other/Mixed | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Bulgaria | 6 | 12 | 9 | 27
  Russia | 129 | 124 | 128 | 381
  Belarus | 7 | 7 | 6 | 20
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] — Population: 1 subject had been mistakenly randomized to the placebo group and was discontinued immediately prior to investigational product administration. Therefore, the patient was included in the ITT population by definition, but no other data except baseline demographics (age, gender, race, ethnicity, and region of inclusion) were collected.
  kg/m^2
    number analyzed (Participants) | 142 | 143 | 142 | 427
    (all) | 26.40 [14.88 to 46.23] | 26.62 [16.98 to 45.52] | 26.93 [17.46 to 51.56] | 26.65 [14.88 to 51.56]
Baseline Disease Severity [Count of Participants; unit: Participants] — The DAS28 (CRP) was calculated using the Swollen joint count (SJC) (28 joints), Tender joint count (TJC) (28 joints), CRP level, and the Patient Global Assessment of Disease Activity Visual Analog Scale (VAS) (100 mm VAS, where 0 is "no disease activity" and 100 was "maximal disease activity") according to the following formula: [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.36 × natural log (CRP+1)] + [0.014 × VAS] + 0.96.
  Participants
    Inactive (DAS28 (CRP) ≤ 3.2) | 0 | 0 | 0 | 0
    Moderately Active (DAS28 (CRP) > 3.2 to ≤ 5.1) | 21 | 18 | 22 | 61
    Very Active (DAS28 (CRP) > 5.1) | 121 | 123 | 119 | 363

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving American College of Rheumatology 20% (ACR20) Response
Description: A responder was defined as any subject satisfying ACR20 criteria and remaining on randomized treatment and in the study at Week 12.
  The calculations were based on a ≥ 20% improvement from baseline in the swollen joint count (SJC) assessed in 66 joints and in the tender joint count (TJC) assessed in 68 joints; and a ≥ 20% improvement from baseline in at least 3 of the 5 remaining core set measures: Patient Global Assessment of Disease Activity (Visual Analog Scale (VAS) assessment), Patient Assessment of Pain (VAS assessment), Health Assessment Questionnaire-Disability Index (HAQ-DI), Physician Global Assessment (VAS assessment), Level of acute phase reactant (CRP or ESR, using level of CRP in this study).
Time Frame: at Week 12
Population: Intent-to-treat (ITT) population: The ITT population includes all randomized subjects. Subjects were analyzed according to the treatment group to which they were randomized. The ITT population is the primary analysis population.
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1: Olokizumab q4w + Methotrexate: Olokizumab 64 mg Subcutaneous q4w + Placebo + Methotrexate (oral)
  Olokizumab 64 mg subcutaneous once every 4 weeks + placebo in order to maintain the blind, subjects randomized to receive OKZ q4w will receive placebo injections at the alternate q4w interval (e.g., Week 2, Week 6, etc.) + concomitant background therapy (Methotrexate) at a stable dose of 15 to 25 mg/week (or ≥10 mg/week if there is documented intolerance to higher doses) with a stable route of administration (oral, subcutaneous, or intramuscular)
- Arm 3: Placebo q2w + Methotrexate: Placebo Subcutaneous q2w + Methotrexate (oral)
  Placebo administered subcutaneously once every 2 weeks + concomitant background therapy (Methotrexate) at a stable dose of 15 to 25 mg/week (or ≥10 mg/week if there is documented intolerance to higher doses) with a stable route of administration (oral, subcutaneous, or intramuscular)
Arm/Group | Arm 1: Olokizumab q4w + Methotrexate | Arm 2: Olokizumab q2w + Methotrexate | Arm 3: Placebo q2w + Methotrexate
Number analyzed (Participants) | 142 | 143 | 143
Participants | 100 | 91 | 37
Statistical Analysis 1: Comparison: Arm 2: Olokizumab q2w + Methotrexate vs Arm 3: Placebo q2w + Methotrexate; The OKZ ACR20 response rates for 64 q2w treatment group at Week 12 are expected to be at least 55%, resulting in an expected difference in ACR20 response rates of 30 percentage points between respective OKZ treatment group and placebo. Sample size yield 100% disjunctive power for testing the primary hypothesis; Test type: Superiority; p < 0.0001, Chi-squared; 2x2 chi-square test; Risk Difference (RD) = 0.378, 97.5% CI 2-sided [0.248 to 0.489]
Statistical Analysis 2: Comparison: Arm 1: Olokizumab q4w + Methotrexate vs Arm 3: Placebo q2w + Methotrexate; The OKZ ACR20 response rates for 64 q4w treatment group at Week 12 are expected to be at least 50%, resulting in an expected difference in ACR20 response rates of 25 percentage points between respective OKZ treatment group and placebo. Sample size yield 100% disjunctive power for testing the primary hypothesis; Test type: Superiority; p < 0.0001, Chi-squared; 2x2 chi-square test; Risk Difference (RD) = 0.445, 97.5% CI 2-sided [0.318 to 0.552]

2. Secondary Outcome: Percentage of Subjects Achieving Low Disease Activity
Description: Defined as Disease Activity Score 28 (DAS28) (CRP) < 3.2, and remaining on randomized treatment and in the study at Week 12.
Time Frame: at Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Arm 3: Placebo q2w + Methotrexate: Placebo Subcutaneous q2w + Methotrexate (oral)
  Placebo administered subcutaneously once every 2 weeks + concomitant background therapy (Methotrexate) at a stable dose of 15 to 25 mg/week (or ≥ 10 mg/week if there is documented intolerance to higher doses) with a stable route of administration (oral, subcutaneous, or intramuscular)
Arm/Group | Arm 1: Olokizumab q4w + Methotrexate | Arm 2: Olokizumab q2w + Methotrexate | Arm 3: Placebo q2w + Methotrexate
Number analyzed (Participants) | 142 | 143 | 143
Participants | 55 | 47 | 5
Statistical Analysis 1: Comparison: Arm 2: Olokizumab q2w + Methotrexate vs Arm 3: Placebo q2w + Methotrexate; DAS28 low disease activity (based on DAS28 [CRP] <3.2) response rate at Week 12 was estimated to be 10% in the placebo group and 30% in 64 q2w OKZ treatment groups respectively, resulting in an expected difference of 20 percentage points between OKZ q2w treatment group and placebo; Test type: Superiority; p < 0.0001, Chi-squared; 2x2 chi-square test; Risk Difference (RD) = 0.294, 97.5% CI 2-sided [0.197 to 0.389]
Statistical Analysis 2: Comparison: Arm 1: Olokizumab q4w + Methotrexate vs Arm 3: Placebo q2w + Methotrexate; DAS28 low disease activity (based on DAS28 [CRP] <3.2) response rate at Week 12 was estimated to be 10% in the placebo group and 22% in 64 mg q4w OKZ treatment group respectively, resulting in an expected difference of 12 percentage points between OKZ q4w treatment group and placebo; Test type: Superiority; p < 0.0001, Chi-squared; 2x2 chi-square test; Risk Difference (RD) = 0.352, 97.5% CI 2-sided [0.251 to 0.449]

3. Secondary Outcome: Improvement of Physical Ability From Baseline to Week 12, as Measured by the Health Assessment Questionnaire Disability Index (HAQ-DI)
Description: Change of physical ability from baseline (the last available assessment prior to the first dose of the study treatment) to week 12, as measured by HAQ-DI. The HAQ-DI total score ranges from 0 (the best outcome) to 3 (the worst outcome).The HAQ-DI assesses the degree of difficulty experienced in 8 domains (dressing and grooming, arising, eating, walking, hygiene, reach, grip, common daily activities) of daily living activities using 20 questions. Each domain consists of 2 or 3 items. For each question the level of difficulty is scored from 0 (without any difficulty, the best outcome) to 3 (unable to do, the worst outcome). Each category is given a score by taking the maximum score of each question. The HAQ-DI was calculated by dividing the sum of the category scores by the number of categories with at least 1 question answered. If fewer than 6 categories had responses, no disability score was calculated.
Time Frame: Baseline to Week 12
Population: Intent-to-treat (ITT) population: The ITT population includes all randomized subjects. Subjects were analyzed according to the treatment group to which they were randomized. The ITT population is the primary analysis population. Subjects with a missing baseline are not included. Data after treatment discontinuation are Included, Data after discontinuing study are multiply Imputed based on the return to baseline assumption.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm 1: Olokizumab q4w + Methotrexate | Arm 2: Olokizumab q2w + Methotrexate | Arm 3: Placebo q2w + Methotrexate
Number analyzed (Participants) | 142 | 141 | 140
score on a scale | -0.52 (0.046) | -0.55 (0.047) | -0.23 (0.044)
Statistical Analysis 1: Comparison: Arm 2: Olokizumab q2w + Methotrexate vs Arm 3: Placebo q2w + Methotrexate; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference = -0.34, 97.5% CI 2-sided [-0.47 to -0.21], Standard Error of Mean 0.059
Statistical Analysis 2: Comparison: Arm 1: Olokizumab q4w + Methotrexate vs Arm 3: Placebo q2w + Methotrexate; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference = -0.36, 97.5% CI 2-sided [-0.49 to -0.23], Standard Error of Mean 0.059

4. Secondary Outcome: Percentage of Subjects Achieving American College of Rheumatology 50% (ACR50) Response
Description: A responder was defined as any subject satisfying ACR50 criteria and remaining on randomized treatment and in the study at Week 24.
  The calculations were based on a ≥ 50% improvement from baseline in the swollen joint count (SJC) assessed in 66 joints and in the tender joint count (TJC) assessed in 68 joints; and a ≥ 50% improvement from baseline in at least 3 of the 5 remaining core set measures: Patient Global Assessment of Disease Activity (Visual Analog Scale (VAS) assessment), Patient Assessment of Pain (VAS assessment), Health Assessment Questionnaire-Disability Index (HAQ-DI), Physician Global Assessment (VAS assessment), Level of acute phase reactant (CRP or ESR, using level of CRP in this study).
Time Frame: at Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1: Olokizumab q4w + Methotrexate: Olokizumab 64 mg Subcutaneous q4w + Placebo + Methotrexate (oral)
  Olokizumab 64 mg Subcutaneous once every 4 weeks+placebo in order to maintain the blind, subjects randomized to receive OKZ q4w will receive placebo injections at the alternate q4w interval (e.g., Week 2, Week 6, etc.) + concomitant background therapy (Methotrexate) at a stable dose of 15 to 25 mg/week (or ≥10 mg/week if there is documented intolerance to higher doses) with a stable route of administration (oral, Subcutaneous, or intramuscular)
Arm/Group | Arm 1: Olokizumab q4w + Methotrexate | Arm 2: Olokizumab q2w + Methotrexate | Arm 3: Placebo q2w + Methotrexate
Number analyzed (Participants) | 142 | 143 | 143
Participants | 69 | 61 | 11
Statistical Analysis 1: Comparison: Arm 2: Olokizumab q2w + Methotrexate vs Arm 3: Placebo q2w + Methotrexate; Test type: Superiority; p < 0.0001, Chi-squared; 2x2 chi-square test; Risk Difference (RD) = 0.350, 97.5% CI 2-sided [0.239 to 0.450]
Statistical Analysis 2: Comparison: Arm 1: Olokizumab q4w + Methotrexate vs Arm 3: Placebo q2w + Methotrexate; Test type: Superiority; p < 0.0001, Chi-squared; 2x2 chi-square test; Risk Difference (RD) = 0.409, 97.5% CI 2-sided [0.296 to 0.509]

5. Secondary Outcome: Percentage of Subjects With Clinical Disease Activity Index (CDAI) ≤ 2.8 (Remission)
Description: Percentage of subjects with Clinical Disease Activity Index (CDAI) ≤ 2.8 (remission) and remaining on randomized treatment and in the study at Week 24
Time Frame: at Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Olokizumab q4w + Methotrexate | Arm 2: Olokizumab q2w + Methotrexate | Arm 3: Placebo q2w + Methotrexate
Number analyzed (Participants) | 142 | 143 | 143
Participants | 11 | 12 | 0
Statistical Analysis 1: Comparison: Arm 2: Olokizumab q2w + Methotrexate vs Arm 3: Placebo q2w + Methotrexate; Test type: Superiority; p < 0.0002, Chi-squared — 2x2 chi-square test; Risk Difference (RD) = 0.084, 97.5% CI 2-sided [0.032 to 0.151]
Statistical Analysis 2: Comparison: Arm 1: Olokizumab q4w + Methotrexate vs Arm 3: Placebo q2w + Methotrexate; Test type: Superiority; p < 0.0003, Chi-squared — 2x2 chi-square test; Risk Difference (RD) = 0.077, 97.5% CI 2-sided [0.027 to 0.143]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from the signature of the informed consent form until the last visit of the subject in the study (up to 22 weeks after the final dose of study treatment) regardless of relationship to study treatment. Any SAE with a start date after the Safety Follow-Up Period was not required to be reported unless the Investigator thought that the event might be related to either the study treatment, study treatment administration, or a protocol procedure.
Description: All AEs and SAEs reported below are related to the Safety Population (safety population included all subjects who receive at least 1 dose of study treatment).
  Data for TEAEs were reported below. A Treatment Emergent Adverse Event (TEAE) is defined as an AE that first occurred or worsened in severity after the first dose of the study treatment.
Arm/Group | Arm 1: Olokizumab q4w + Methotrexate | Arm 2: Olokizumab q2w + Methotrexate | Arm 3: Placebo q2w + Methotrexate
All-Cause Mortality (participants affected / at risk) | 0/142 | 1/143 | 0/142
Serious Adverse Events (participants affected / at risk) | 8/142 | 8/143 | 4/142
Other Adverse Events (participants affected / at risk) | 53/142 | 51/143 | 35/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Olokizumab q4w + Methotrexate (N=142) | Arm 2: Olokizumab q2w + Methotrexate (N=143) | Arm 3: Placebo q2w + Methotrexate (N=142)
Alanine aminotransferase increased (Investigations) | 4 (5) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Toxic shock syndrome (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cervix carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic vascular disorder (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Olokizumab q4w + Methotrexate (N=142) | Arm 2: Olokizumab q2w + Methotrexate (N=143) | Arm 3: Placebo q2w + Methotrexate (N=142)
Alanine aminotransferase increased (Investigations) | 30 (44) | 25 (32) | 11 (14)
Aspartate aminotransferase increased (Investigations) | 19 (27) | 16 (22) | 10 (12)
White blood cell count decreased (Investigations) | 6 (13) | 7 (9) | 4 (5)
Neutrophil count decreased (Investigations) | 7 (10) | 6 (6) | 3 (4)
Nasopharyngitis (Infections and infestations) | 3 (3) | 4 (4) | 6 (8)
Upper respiratory tract infection (Infections and infestations) | 6 (9) | 2 (2) | 4 (4)
Blood cholesterol increased (Investigations) | 4 (4) | 6 (7) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 7 (10) | 8 (10) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 9 (11) | 5 (6) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 4 (4) | 6 (9)
Gamma-glutamyltransferase increased (Investigations) | 6 (9) | 3 (5) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study related information could be made public available only after Sponsors written permission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-30): https://cdn.clinicaltrials.gov/large-docs/68/NCT02760368/Prot_SAP_000.pdf